CLINICAL TRIAL: NCT01979523
Title: A Randomized Two-Arm Phase II Study of Trametinib Alone and in Combination With GSK2141795 in Patients With Advanced Uveal Melanoma
Brief Title: Trametinib With or Without GSK2141795 in Treating Patients With Metastatic Uveal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02091; NCI-2013-02091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-144; 9445 (Other: Memorial Sloan Kettering Cancer Center); 9445 (Other: CTEP); N01CM00039 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Uveal Melanoma; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — trametinib; omipalisib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience objective disease progression may crossover to Arm B. (no patients will be enrolled to Arm B or Crossover therapy as of 11/6/2015)
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Trametinib
- Arm B (trametinib, Akt inhibitor GSK2141795) (Experimental): Patients receive trametinib PO QD and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Trametinib; Drug: Uprosertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212
Drug: Uprosertib — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795
  Arms: Arm B (trametinib, Akt inhibitor GSK2141795)

SUMMARY:
This randomized phase II trial studies how well trametinib with or without Akt inhibitor GSK2141795 (GSK2141795) works in treating patients with uveal melanoma that has spread to other parts of the body (metastatic). Trametinib and GSK2141795 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether trametinib is more effective with or without GSK2141795 in treating patients with metastatic uveal melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival between those treated with trametinib alone and those treated with the combination of trametinib and GSK2141795.

SECONDARY OBJECTIVES:

I. To compare overall survival between those treated with trametinib alone and those treated with the combination of trametinib and GSK2141795.

II. To compare the overall response rate between those treated with trametinib alone and those treated with the combination of trametinib and GSK2141795.

III. To compare the safety and toxicity between those treated with trametinib alone and those treated with the combination of trametinib and GSK2141795.

EXPLORATORY OBJECTIVES:

I. To assess clinical outcomes (response rate, progression-free and overall survival) with trametinib and GSK2141795 after progression on trametinib.

II. To assess toxicity with trametinib and GSK2141795 after progression on trametinib.

III. To correlate clinical outcome with Gnaq/11 mutational status. IV. To assess the pharmacodynamic effects of trametinib alone and with GSK2141795, and utilize whole-transcriptome and reverse phase protein array to identify markers of sensitivity and primary resistance to trametinib alone and with GSK2141795.

V. To assess for changes in circulating tumor deoxyribonucleic acid (DNA) with therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience objective disease progression may crossover to Arm B. (no patients will be enrolled to Arm B or Crossover therapy as of 11/6/2015)

ARM B: Patients receive trametinib PO QD and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic histologically or cytologically confirmed uveal melanoma; if histologic or cytologic confirmation of the primary is not available, confirmation of the primary diagnosis of uveal melanoma by the treating investigator can be clinically obtained, as per standard practice for uveal melanoma; pathologic confirmation of metastatic disease will be performed at Memorial Sloan Kettering (MSK) or at a participating site
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients may not have received prior systemic or hepatic directed infusional/embolization therapies for advanced uveal melanoma; local therapies such as radiofrequency ablation or cryotherapy for metastatic disease are permitted but must have been performed at least 21 days prior to initiation of study therapy; lesions treated with local modalities such as radiofrequency ablation or cryotherapy may not be used as target lesions unless they demonstrate growth over a minimum of 3 months on subsequent imaging studies
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version (v)4 grade =< 1 (except alopecia) at the time of randomization and crossover
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL (not requiring transfusions within the past 2 weeks)
* Total bilirubin =< 1.5 x institutional upper limit of normal; Note: patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal for patients with no concurrent liver metastases, OR =< 2.5 x institutional upper limit of normal for patients with concurrent liver metastases
* Creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative blood pregnancy test within 14 days prior to start of protocol treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients must agree to provide all imaging studies for central radiology review; this central radiology review may be performed retrospectively and will not be utilized for decision making for patients on study
* ELIGIBILITY CRITERIA FOR CROSSOVER REGISTRATION
* Previously treated with trametinib on Arm A and experienced objective disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Not removed from trametinib treatment due to the development of unacceptable toxicity that is not manageable with dose reduction
* No other drug treatment for malignant melanoma administered after completing study treatment with trametinib
* Meet all eligibility criteria with the exception of:

  * Prior therapy with trametinib will be permitted
  * All laboratory parameters must be met as outlined except for ALT and total bilirubin, which must meet criteria for continued therapy
  * Patients who are eligible for cross-over will not need to undergo another ophthalmologic examination

Exclusion Criteria:

* History of another malignancy except for those who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies not requiring active therapy, are eligible; consult the study MSK Principal Investigator or the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Any major surgery or extensive radiotherapy within 21 days prior to randomization and crossover
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib alone or with GSK2141795 and during the study
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression; treated brain metastases must have been stable for at least 1 month
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, GSK2141795, or excipients or to dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication
* History or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED) in the eye unaffected by uveal melanoma
* Patients with abnormal fasting glucose values (values > upper limit of normal [ULN] or < LLN) at screening will be excluded; in addition, patients with type 1 diabetes will also be excluded; however, patients with type 2 diabetes will be allowed if diagnosed >= 6 months prior to enrollment, and if presenting with a normal fasting glucose value and a regular hemoglobin A1C (HbA1C) =< 8% at screening
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricular ejection fraction (LVEF) < LLN
  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2026-07-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Shoushtari, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (5):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
- Institut Curie Paris, Paris, France
- The University of Liverpool, Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795) | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Full Range); unit: years] | 59 [32 to 74] | 59.6 [24 to 74] | 59.3 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (Progression-free Survival [PFS]), Defined From the Date of Randomization to the Date of Documented Progression or Death Per RECIST
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from randomization to the earlier date of objective disease progression or death
Population: This assessment corresponds to the participants' initial treatment assignment.
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 20 | 21
weeks | 16.6 [3.3 to 43.7] | 15.6 [3.9 to 137]
Statistical Analysis 1: Comparison: Arm A (Trametinib) vs Arm B (Trametinib, Akt Inhibitor GSK2141795); Test type: Other; p = 0.74, Log Rank

2. Secondary Outcome: Number of Participants With Toxicity, Graded According to the National Cancer Institute CTCAE v4.0, Who Were Treated and Did Not Withdraw Consent
Description: Graded according to the National Cancer Institute CTCAE v4.0. Please see AE/SAE Section for specifics.
Time Frame: From date of randomization until the date of death from any cause or 4 weeks from last treatment of the initial treatment assignment, whichever came first, assessed up to 12 months
Population: This assessment corresponds to the participants' initial treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 21 | 21
Participants | 21 | 21

3. Secondary Outcome: Overall Survival (OS) Per RECIST Criteria
Description: OS curves will be generated using Kaplan-Meier methodology.
Time Frame: up to 36 months
Population: This assessment corresponds to the participants' initial treatment assignment.
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 20 | 21
weeks | 69 [3.3 to 139] | 88 [4.1 to 152]

4. Secondary Outcome: Response Rate (Complete Response+ Partial Response) Using the RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: as for outcome 2
Population: This assessment corresponds to the participants' initial treatment assignment.
Measure: Number; unit: participants
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 19 | 18
participants
  Partial Response | 2 | 1
  Progression of Disease | 8 | 4
  Stable Disease | 9 | 13

5. Other Pre Specified Outcome: Change in Apoptosis in Paired Samples as Assessed by Caspase 3 Cleavage
Time Frame: Baseline to 4 weeks from last treatment
Population: The size of the cores from the acquired samples in almost all participants were small and the quality was insufficient to analyze across the sample set.
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Change in Suppression of Phosphorylated (p)-ERK, AKT, and Cyclin-D1
Description: Association between suppression and response to treatment will be assessed using Fisher's exact test.
Time Frame: Baseline to 4 weeks from last treatment
Population: as for outcome 5
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Circulating Tumor DNA Levels
Description: The numeric data will be summarized by clinical response.
Time Frame: Up to 4 weeks from last treatment
Population: Data were not analyzed due to lack of funding.
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Gnaq/11 Mutational Status
Description: Clinical response will be associated with Gnaq/11 mutational status using Wilcoxon rank sum test.
Time Frame: Up to 4 weeks from last treatment
Population: Analysis across the sample set unable to be completed due to patient-specific issues (participants skipped biopsy for safety, insufficient cores for extra DNA extraction)
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of death from any cause or 4 weeks from removal of the study, whichever came first, assessed up to 12 months
Description: AE's and SAE's for Arm A, Arm B, and the crossover group were collected.
Groups:
- Crossover Arm: Participants had progression of disease on Arm A and were then treated on Arm B.
Arm/Group | Arm A (Trametinib) | Arm B (Trametinib, Akt Inhibitor GSK2141795) | Crossover Arm
All-Cause Mortality (participants affected / at risk) | 5/20 | 13/21 | 8/11
Serious Adverse Events (participants affected / at risk) | 8/20 | 12/21 | 11/11
Other Adverse Events (participants affected / at risk) | 20/20 | 21/21 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Trametinib) (N=20) | Arm B (Trametinib, Akt Inhibitor GSK2141795) (N=21) | Crossover Arm (N=11)
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Edema face (General disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Retinal vascular disorder (Eye disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Endocarditis infective (Infections and infestations) | 0 | 1 | 0
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 3 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 1 | 9
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Trametinib) (N=20) | Arm B (Trametinib, Akt Inhibitor GSK2141795) (N=21) | Crossover Arm (N=11)
Alanine aminotransferase increased (Investigations) | 0 | 5 | 5
Alkaline phosphatase increased (Investigations) | 3 | 6 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 7 | 0
Blood bilirubin increased (Investigations) | 3 | 3 | 0
Blurred vision (Eye disorders) | 2 | 0 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0
CPK increased (Investigations) | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 6
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 2
Ejection fraction decreased (Investigations) | 4 | 1 | 0
Fatigue (General disorders) | 0 | 6 | 6
Headache (Nervous system disorders) | 1 | 2 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 4
Hypertension (Vascular disorders) | 4 | 10 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2 | 0
INR increased (Investigations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 5
Musculoskeletal & conn tissue disorder Other, spec (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 6
Neutrophil count decreased (Investigations) | 2 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4 | 6
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin infection (Infections and infestations) | 2 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 4
White blood cell decreased (Investigations) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Edema trunk (General disorders) | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Vulval infection (Infections and infestations) | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 5
Weight loss (Investigations) | 0 | 0 | 4
WBC Decreased (Investigations) | 0 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT01979523/Prot_SAP_000.pdf